CLINICAL TRIAL: NCT05517057
Title: Assessment of a Predictive Radiologic Score to Predict the Failure of the Non-operative Management of Adhesive Small Bowel Obstruction: a Prospective Cohort Analysis
Brief Title: Radiologic Score and Failure of Conservative Management of Adhesive Small Bowel Obstruction
Acronym: PREDIFAIL
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-099
Record Dates: First submitted 2022-08-20; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Small Bowel Obstruction; Conservative Management; Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- success of the medical management: Patients that recovered flatus and stools, and that tolerated solid food within the 3 days after the admission
- failure of the medical management: Patients that did not recover flatus and stools, and that did not tolerate solid food within the 3 days after the admission. These patients had an indication for surgery.

SUMMARY:
The management of acute adhesive small bowel obstruction remains challenging for the digestive surgeon. The Bologna guidelines recommend that conservative management of aSBO. The literature reports that this form of management has a failure rate between 10 and 40%.

A radiological score has been proposed and was associated with an increased risk of failure of conservative management.

This tool is promising to select patients further requiring surgery but it has to be assessed in a multi centric prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* all the consecutive patients admitted for initial non-surgical management for aSBO
* during the period of inclusion

Exclusion Criteria:

* the cause of SBO was functional or other than adhesive
* patients requiring initial surgical management.
* absence of computed tomography performed at admission

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was an observational multicentric cohort study including all the consecutive patients admitted for initial non-surgical management for aSBO. The study took place over a period of 3 months (September 15 - December 15, 2021) in 15 French centers.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Angers CT score | immediately after the completion of the CT-scan
  The Angers CT score ≥5 was considered to be risk factor for failure of the medical management.
  Angers CT score was calculated by reading the CT scan as follow:
  * beak sign (+2), if not (0)
  * closed loop (+4), if not (0)
  * focal (+4) or diffuse (+4) intraperitoneal liquid, if not (0)
  * focal (+2) or diffuse (0) mesenteric haziness, if not (0)
  * focal (-3) or diffuse (-3) mesenteric liquid, if not (0)
  * diameter of the most dilated small bowel loop > 40 mm (-2) (if not (0).

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital of Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No